CLINICAL TRIAL: NCT06579534
Title: Exploring the Effectiveness of Multimedia Health Education Guidance on Risk Perception, Self-Health Management, and Fall Prevention Among Frail Patients
Brief Title: Multimedia Education for Frail Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AsiaU1
Record Dates: First submitted 2024-07-27; First posted 2024-08-30 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-08

CONDITIONS: Frailty
Keywords: Fall; Frailty; Multimedia Health Education
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: Control and Experimental group
Who Masked: Participant
Masking Description: Fall prevention education before discharge is an inevitable measure. Participants accepted such measures but did not know that this study involved differentiated health education methods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Device: Oral Explanation of Paper-Based Health Education (No Intervention): Before the patient is discharged from the hospital, the nurse orally informs the patient about the precautions for preventing falls after discharge using a discharge health education leaflet.
- Device: Multimedia Video Health Education on Fall Prevention (Experimental): Multimedia audio-visual health education tools: Taking fall risk factors, self-health management and fall prevention measures as the main teaching plan, investigators produce multimedia digital audio-visual teaching materials in Chinese version for adults, Chinese version for children, and English version for adults, with built-in AI patented artificial intelligence automatic dubbing, and matching Chinese or English subtitles and lively 3D virtual lecturers are presented on the screen to explain the course, and pictures, physical photos, short videos, etc. are used as the main content, allowing viewers to quickly and conveniently grasp the key points and absorb knowledge.
  Interventions: Other: Health education strategy

INTERVENTIONS:
Other: Health education strategy — Based on the concept of precise health care, investigators design risk awareness, self-health management and fall prevention care measures, and provide inpatients with high-risk groups with frailty and falls with health education guidance on muscle endurance training and fall prevention. This study adopts purposive sampling, randomization, assignment, and parallel experiments to divide into a control group and an experimental group. The control group uses conventional health education guidance to provide fall prevention education, and the experimental group uses multimedia health education videos to provide education to patients or primary caregivers. Provide health education on the risk, management and prevention of falls.
  Arms: Device: Multimedia Video Health Education on Fall Prevention

SUMMARY:
The goal of this clinical trial is to explore the impact of precision health care interventions on inpatients in acute medical institutions regarding their risk of falls, management, and prevention knowledge, as well as the incidence of falls among these patients. The main questions it aims to answer are:

What is the effectiveness of precision health care interventions on inpatients' knowledge of fall risk in acute medical institutions? What is the effectiveness of precision health care interventions on inpatients' knowledge of fall management in acute medical institutions? What is the effectiveness of precision health care interventions on inpatients' knowledge of fall prevention in acute medical institutions?

DETAILED DESCRIPTION:
Frailty relates to the concept of physical deterioration associated with the aging process, which includes a weakening of the physiological and integrated physical strength of the body, its reserve and resistance to stressors, resulting in poor health, such as loss of physical and mental performance. Frailty is an important health care topic in patients with geriatric syndromes. Once the elderly enter the early stage of frailty, they are likely to fall repeatedly. Studies have shown that frailty and premature aging are important predictors of falls in the elderly. Therefore, professional medical staff should use frailty assessment indicators as early as possible to assess the possibility of frailty among the elderly in medical institutions or communities. At the same time, effective prevention strategies should be adopted to prevent reduce the incidence of falls due to frailty and improve the quality of life of patients and the elderly. Therefore, assessment of possible falls and frailty risks is a priority in acute care settings.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted to general acute wards and surgical patients
2. Fall assessment score ≥ 3% of the high-risk group for falls

Exclusion Criteria:

1. Patients who were bedridden for a long time before admission
2. Patients suffering from mental illness
3. The patient or primary caregiver cannot respond effectively

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
inpatients' knowledge of fall risk in acute medical institutions | discharge day (assessed up to 1 days)
  Fall Risk Assessment Scale:
  Knowledge related to fall risk is a self-compiled questionnaire with a total of 5 questions. The estimated test time is 3 to 5 minutes.
  Answer with true or false questions, each question is worth 20 points, and the score ranges from 0 to 100 points.
  The higher the score, the better the knowledge level.
inpatients' knowledge of fall management in acute medical institutions | discharge day (assessed up to 1 days)
  Fall Prevention Self-health Management Scale:
  The knowledge related to fall prevention and self-health management is a self-constructed questionnaire with a total of 5 questions. The estimated test time is 3 to 5 minutes.
  Answer with true or false questions, each question is worth 20 points, and the score ranges from 0 to 100 points.
  The higher the score, the better the knowledge level.
inpatients' knowledge of fall prevention in acute medical institutions | discharge day (assessed up to 1 days)
  Fall Prevention Scale Knowledge related to fall prevention is a self-constructed questionnaire with a total of 5 questions.
  Answer with true or false questions, each question is worth 20 points, and the score ranges from 0 to 100 points.
  The higher the score, the better the knowledge level.

CONTACTS AND LOCATIONS:
Overall Officials: Hua-Shan Wu, Study Chair — Asia University

IPD SHARING:
Plan to Share IPD: No